CLINICAL TRIAL: NCT01171963
Title: Efficacy, Immunogenicity and Safety of Two Doses of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Liquid Human Rotavirus (HRV) Vaccine (444563), in Healthy Infants
Brief Title: Study to Assess the Efficacy, Immunogenicity and Safety of Liquid Human Rotavirus Vaccine, in Healthy Chinese Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 113808
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-06

CONDITIONS: Infections, Rotavirus
Keywords: Liquid human retrovirus vaccine
MeSH Terms: conditions — Rotavirus Infections | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Pentetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rotarix Group (Experimental): Subjects aged between and including 6 and 16 weeks at the time of first vaccination received 2 doses of Rotarix™ vaccine, liquid formulation, at Day 0 and at Month 1. As part of the routine childhood vaccination according to the Expanded Program of Immunization (EPI) recommendations in China, subjects in this group also received 3 doses of Infanrix™ vaccine and 3 doses of the oral poliovirus vaccine manufactured by the Institute of Medical Biology of the Chinese Academy of Medical Sciences (OPV). The Infanrix™ and the OPV vaccines were administered independently of (Sub-cohort 1) or concomitantly with (Sub-cohort 2) the Rotarix™ vaccine. When administered concomitantly, subjects received the 3 doses of Infanrix™ vaccine at Months 1, 2 and 3, and the 3 doses of the OPV vaccine at Day 0, Month 1 and Month 2. The Rotarix™ and OPV vaccines were administered orally; the Infanrix™ vaccine was administered intramuscularly in the left anterolateral thigh.
  Interventions: Biological: GSK Biologicals' liquid human rotavirus vaccine 444563; Biological: Infanrix™; Biological: Institute of Medical Biology Chinese Academy of Medical Sciences' Oral poliovirus vaccine (OPV)
- Placebo Group (Placebo Comparator): Subjects aged between and including 6 and 16 weeks at the time of first vaccination received 2 doses of Placebo at Day 0 and at Month 1. As part of the routine childhood vaccination according to the Expanded Program of Immunization (EPI) recommendations in China, subjects in this group also received 3 doses of Infanrix™ vaccine and 3 doses of the oral poliovirus vaccine manufactured by the Institute of Medical Biology of the Chinese Academy of Medical Sciences (OPV). The Infanrix™ and the OPV vaccine were administered independently of (Sub-cohort 1) or concomitantly with (Sub-cohort 2) the Placebo. When administered concomitantly, subjects received the 3 doses of Infanrix™ vaccine at Months 1, 2 and 3, and the 3 doses of the OPV vaccine at Day 0, Month 1 and Month 2. The Placebo and the OPV vaccine were administered orally; the Infanrix™ vaccine was administered intramuscularly in the left anterolateral thigh.
  Interventions: Biological: Placebo; Biological: Infanrix™; Biological: Institute of Medical Biology Chinese Academy of Medical Sciences' Oral poliovirus vaccine (OPV)

INTERVENTIONS:
Biological: GSK Biologicals' liquid human rotavirus vaccine 444563 — Oral administration
  Arms: Rotarix Group
Biological: Placebo — Oral administration
  Arms: Placebo Group
Biological: Infanrix™ — Intramuscular administration
  Other Names: DTPa
Biological: Institute of Medical Biology Chinese Academy of Medical Sciences' Oral poliovirus vaccine (OPV) — Oral administration

SUMMARY:
The purpose of this study is to assess the efficacy, immunogenicity and safety of GSK Biologicals' liquid human rotavirus vaccine in healthy Chinese infants 6 to 16 weeks of age.

DETAILED DESCRIPTION:
Subjects can receive routine childhood vaccination according to the expanded program of immunisation recommendations in China.

There will be two treatment groups (liquid human rotavirus vaccine and placebo). The study will also have two immunogenicity subgroups comprising of few subjects from both the treatment groups. The immunogenicity subgroup 1 will assess the immunogenicity of the liquid human rotavirus vaccine and the immunogenicity subgroup 2 will assess the immunogenicity of liquid human rotavirus vaccine and also the immunogenicity of oral poliovirus vaccine and diphtheria tetanus and acellular pertussis vaccine given concomitantly with liquid human rotavirus vaccine or placebo.

This protocol posting has been updated following the Protocol Amendment 2, dated 05 August 2011. The impacted section in the protocol posting is: Outcome Measures Section.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/Legally Acceptable Representatives can and will comply with the requirements of the protocol.
* A male or female infant of Chinese origin between, and including, 6 and 16 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parents/Legally Acceptable Representatives of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 14 days before each dose of study vaccine(s) and ending 14 days after the first dose of the human rotavirus vaccine or placebo except for the routine childhood vaccinations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any clinically significant history of gastrointestinal disease including any uncorrected congenital malformation (such as Meckel's diverticulum) of the gastrointestinal tract that would predispose for intussusception .
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of confirmed rotavirus gastroenteritis.
* Acute disease and/or fever at the time of enrolment.
* Gastroenteritis within 7 days preceding the study vaccine or placebo administration.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

In addition to the criteria mentioned above, the following criteria will be applicable to all subjects in the immunogenicity subgroup 2:

* History of diphtheria, tetanus and pertussis disease.
* History of seizures or progressive neurological disease.
* Previous vaccination against diphtheria, tetanus, pertussis and poliomyelitis.

Ages: 6 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3340 (Actual)
Dates: Start 2010-08-29; Primary Completion 2012-05-12 (Actual); Study Completion 2012-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- China (4):
  - GSK Investigational Site, Hechi, Guangxi
  - GSK Investigational Site, Liucheng County, Guangxi
  - GSK Investigational Site, Liuchow, Guangxi
  - GSK Investigational Site, Luzhai County, Guangxi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Li RC, Huang T, Li Y, Luo D, Tao J, Fu B, Si G, Nong Y, Mo Z, Liao X, Luan I, Tang H, Rathi N, Karkada N, Han HH. Human rotavirus vaccine (RIX4414) efficacy in the first two years of life: a randomized, placebo-controlled trial in China. Hum Vaccin Immunother. 2014;10(1):11-8. doi: 10.4161/hv.26319. Epub 2013 Sep 6. PMID 24013441
- [Derived] Li RC, Li YP, Mo ZJ, Luo D, Huang T, Kong JL, Wang LH, Song NS, Liu A, Zhang H, Liao X, Karkada N, Han HH. Reactogenicity and safety of a liquid human rotavirus vaccine (RIX4414) in healthy adults, children and infants in China: randomized, double-blind, placebo-controlled Phase I studies. Hum Vaccin Immunother. 2013 Aug;9(8):1638-42. doi: 10.4161/hv.25076. Epub 2013 Jun 4. PMID 23807360
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Duration of the study was of a maximum of 21 months, with the enrolment of subjects starting in August 2010, and subjects being followed up to May 2012 (study Month 21 and Study End), end of the rotavirus season in China.
Pre-assignment Details: Subjects were assigned to 2 sub-cohorts (1:1 ratio). Sub-cohort 1 and Sub-cohort 2 subjects received their OPV and Infanrix™ EPI vaccination respectively independently of, and concomitantly with their Rotarix™/placebo vaccination. 3340 subjects were allocated study subject number allocated and 3333 vaccinated .
Period: Overall Study
Arm/Group | Rotarix Group | Placebo Group
Started | 1666 | 1667
Completed | 1518 | 1499
Not Completed | 148 | 168
Not completed — Adverse Event | 10 | 15
Not completed — Lost to Follow-up | 23 | 24
Not completed — Other - diarrhoea | 1 | 0
Not completed — Withdrawal by Subject | 114 | 129

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 1666 | 1667 | 3333
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.5 (2.64) | 9.7 (2.59) | 9.6 (2.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 795 | 836 | 1631
  Male | 871 | 831 | 1702

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Severe Episode(s) of Rotavirus Gastroenteritis (RVGE) Caused by the Circulating Wild Type (WT) Strains
Description: A gastroenteritis episode was classified positive for rotavirus (RV) and caused by the circulating wild-type (WT) RV strains if RV other than the vaccine strain was identified in a stool sample collected during the episode. Severe RVGE was defined as an episode of RV GE with score equal to or higher than (>=) 11 on a 20-point Vesikari scoring system.
Time Frame: From Month 1 ½ to Month 21
Population: The analysis was performed on the According-to-Protocol cohort for efficacy, which included subjects vaccinated with Rotarix™ vaccine or placebo who had entered the efficacy surveillance period (Months 1 ½-21) with no rotavirus other than vaccine strain in the gastroenteritis stool samples collected between Day 0 and Month 1 ½.
Measure: Count of Participants; unit: Participants
Groups:
- Rotarix Group: Subjects aged between and including 6 and 16 weeks at the time of first vaccination received 2 doses of Rotarix vaccine, liquid formulation, at Day 0 and at Month 1. As part of the routine childhood vaccination according to the Expanded Program of Immunization (EPI) recommendations in China, subjects in this group also received 3 doses of Infanrix vaccine and 3 doses of the oral poliovirus vaccine manufactured by the Institute of Medical Biology of the Chinese Academy of Medical Sciences (OPV). The Infanrix and the OPV vaccines were administered independently of (Sub-cohort 1) or concomitantly with (Sub-cohort 2) the Rotarix vaccine. When administered concomitantly, subjects received the 3 doses of Infanrix vaccine at Months 1, 2 and 3, and the 3 doses of the OPV vaccine at Day 0, Month 1 and Month 2. The Rotarix and OPV vaccines were administered orally; the Infanrix vaccine was administered intramuscularly in the left anterolateral thigh.
- Placebo Group: Subjects aged between and including 6 and 16 weeks at the time of first vaccination received 2 doses of Placebo at Day 0 and at Month 1. As part of the routine childhood vaccination according to the Expanded Program of Immunization (EPI) recommendations in China, subjects in this group also received 3 doses of Infanrix vaccine and 3 doses of the oral poliovirus vaccine manufactured by the Institute of Medical Biology of the Chinese Academy of Medical Sciences (OPV). The Infanrix and the OPV vaccine were administered independently of (Sub-cohort 1) or concomitantly with (Sub-cohort 2) the Placebo. When administered concomitantly, subjects received the 3 doses of Infanrix vaccine at Months 1, 2 and 3, and the 3 doses of the OPV vaccine at Day 0, Month 1 and Month 2. The Placebo and the OPV vaccine were administered orally; the Infanrix vaccine was administered intramuscularly in the left anterolateral thigh.
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1575 | 1573
Participants | 21 | 75

2. Secondary Outcome: Number of Subjects With Any Episode(s) of Rotavirus Gastroenteritis (RVGE) Caused by the Circulating Wild-type Strains
Description: A gastroenteritis episode was classified positive for rotavirus (RV) and caused by the circulating wild-type (WT) RV strains if RV other than the vaccine strain was identified in a stool sample collected during the episode.
Time Frame: From Month 1 ½ to Month 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1575 | 1573
Participants | 70 | 167

3. Secondary Outcome: Number of Subjects With Any Episode(s) of Rotavirus Gastroenteritis (RVGE) of Any Type.
Description: A gastroenteritis episode was classified positive for rotavirus (RV) if RV was identified in a stool sample collected during the episode. RV types assessed were G1 Wild Type (G1WT), G2, G3, G9, GX (G type unknown, but not vaccine strain), P4, P8 Wild Type (P8WT), P9, PX (P type unknown, but not vaccine strain) and Pooled Non-G1WT.
Time Frame: From Month 1 ½ to Month 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1575 | 1573
Participants
  Subjects with G1WT RVGE | 22 | 46
  Subjects with G2 RVGE | 42 | 105
  Subjects with G3 RVGE | 1 | 12
  Subjects with G9 RVGE | 1 | 5
  Subjects with GX RVGE | 6 | 8
  Subjects with P4 RVGE | 43 | 107
  Subjects with P8WT RVGE | 25 | 59
  Subjects with P9 RVGE | 0 | 1
  Subjects with PX RVGE | 4 | 1
  Subjects with Pooled Non-G1WT RVGE | 49 | 129

4. Secondary Outcome: Number of Subjects With Severe Episode(s) of Rotavirus Gastroenteritis (RVGE) of Any Type.
Description: A gastroenteritis episode was classified positive for rotavirus (RV) if RV was identified in a stool sample collected during the episode. Severe RVGE was defined as an episode of RVGE with score equal to or higher than (>=) 11 on a 20-point Vesikari scoring system. RV types assessed were G1 Wild Type (G1WT), G2, G3, G9, GX (G type unknown, but not vaccine strain), P4, P8 Wild Type (P8WT), P9, PX (P type unknown, but not vaccine strain) and Pooled Non-G1WT.
Time Frame: From Month 1 ½ to Month 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Rotarix Group: Subjects aged between and including 6 and 16 weeks at the time of first vaccination received 2 doses of Rotarix vaccine, liquid formulation, at Day 0 and at Month 1. As part of the routine childhood vaccination according to the Expanded Program of Immunization (EPI) recommendations in China, subjects in this group also received 3 doses of Infanrix vaccine and 3 doses of the oral poliovirus vaccine manufactured by the Institute of Medical Biology of the Chinese Academy of Medical Sciences (OPV). The Infanrix and the OPV vaccines were administered independently of (Sub-cohort 1) or concomitantly with (Sub-cohort 2) the Rotarix vaccine. When administered concomitantly, subjects received the 3 doses of Infanrix vaccine at Months 1, 2 and 3, and the 3 doses of the OPV vaccine at Day 0, Month 1 and Month 2. The Rotarix and OPV vaccines were administered orally; the Infanrix vaccine was administered intramuscularly in the left anterolateral thigh.Not Applicable
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1575 | 1573
Participants
  Subjects with severe G1WT RVGE | 9 | 25
  Subjects with severe G2 RVGE | 11 | 43
  Subjects with severe G3 RVGE | 0 | 3
  Subjects with severe G9 RVGE | 0 | 3
  Subjects with severe GX RVGE | 1 | 6
  Subjects with severe P4 RVGE | 12 | 43
  Subjects with severe P8WT RVGE | 9 | 31
  Subjects with severe PX RVGE | 1 | 1
  Subjects with severe Pooled Non-G1WT RVGE | 12 | 54

5. Secondary Outcome: Number of Subjects With Episodes of Rotavirus Gastroenteritis (RVGE) Caused by the Circulating Wild Type (WT) Strains Requiring Hospitalization
Description: A gastroenteritis episode was classified positive for rotavirus (RV) and caused by the circulating WT RV strains if RV other than the vaccine strain was identified in a stool sample collected during the episode.
Time Frame: From Month 1 ½ to Month 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1575 | 1573
Participants | 4 | 21

6. Secondary Outcome: Number of Subjects With Any and Severe Gastroenteritis (GE) Due to Any Cause
Description: Severe GE was defined as an episode of GE with score equal to or higher than (>=) 11 on a 20-point Vesikari scoring system. This outcome measure concerns results for GE episodes due to any cause.
Time Frame: From Month 1 ½ to Month 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1575 | 1573
Participants
  Subjects with any GE | 728 | 759
  Subjects with any severe GE | 187 | 206

7. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms Following Vaccination With the Rotarix Vaccine/Placebo
Description: Assessed solicited general symptoms were fever,defined as axillary temperature (T) above or equal to [>=] 37.5 degrees Celsius [°C] (if GSK scale) or >= 37.1°C (if Chinese scale), fussiness/irritability, loss of appetite, cough/runny nose, diarrhea and vomiting. Any = any occurrence of the specified solicited general symptom regardless of the intensity grade or relationship to vaccination. This outcome measure was only assessed in subjects from Sub-cohort 1, who received the EPI vaccination independently of study vaccination with the Rotarix vaccine/placebo.
Time Frame: Within the 8-day (Days 0-7) follow-up periods after any dose of Rotarix vaccine/placebo
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented, solely on subjects not part of Sub-cohort 2.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Group: Subjects aged between and including 6 and 16 weeks at the time of first vaccination received 2 doses of Placebo at Day 0 and at Month 1. As part of the routine childhood vaccination according to the Expanded Program of Immunization (EPI) recommendations in China, subjects in this group also received 3 doses of Infanrix vaccine and 3 doses of the oral poliovirus vaccine manufactured by the Institute of Medical Biology of the Chinese Academy of Medical Sciences (OPV). The Infanrix and the OPV vaccine were administered independently of (Sub-cohort 1) or concomitantly with (Sub-cohort 2) the Placebo. When administered concomitantly, subjects received the 3 doses of Infanrix™ vaccine at Months 1, 2 and 3, and the 3 doses of the OPV vaccine at Day 0, Month 1 and Month 2. The Placebo and the OPV vaccine were administered orally; the Infanrix vaccine was administered intramuscularly in the left anterolateral thigh.
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1513 | 1514
Participants
  Any cough/runny nose | 313 | 366
  Any diarrhoea | 127 | 123
  Any Irritability/Fussiness | 415 | 448
  Any Loss of appetite | 253 | 250
  Any Fever - Chinese scale: Axillary T >= 37.1°C | 302 | 313
  Any Fever - GSK scale: Axillary T >= 37.5°C | 83 | 104
  Any Vomiting | 213 | 232

8. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms Following Administration of the Co-administered EPI Vaccines
Description: Solicited general symptoms assessed following administration of the co-administered EPI vaccines were drowsiness, gastrointestinal symptoms, fussiness/irritability, loss of appetite, and fever, defined as axillary temperature (T) above or equal to [>=] 37.5 degrees Celsius [°C] (if GSK scale) or >= 37.1°C (if Chinese scale ). Any = any occurrence of the specified solicited general symptom regardless of the intensity grade or relationship to vaccination. This outcome measure was only assessed in subjects from Sub-cohort 2, who received the EPI vaccination concomitantly with study vaccination with the Rotarix vaccine/placebo.
Time Frame: Within the 8-day (Days 0-7) follow-up periods following Doses 1 and 2 of the OPV vaccine and Dose 1 of the Infanrix vaccine
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 153 | 153
Participants
  Any Drowsiness | 44 | 38
  Any Gastrointestinal symptoms | 43 | 38
  Any Irritability/Fussiness | 56 | 52
  Any Loss of appetite | 43 | 32
  Any Fever - Chinese scale: Axillary T >= 37.1°C | 18 | 20
  Any Fever - GSK scale: Axillary T >= 37.5°C | 6 | 7

9. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms Following Dose 2 of the Rotarix Vaccine/Placebo
Description: Solicited local symptoms assessed following administration of the co-administered EPI vaccines were pain, swelling, and redness. Any = any occurrence of the specified solicited local symptom regardless of the intensity grade. This outcome measure was only assessed in subjects from Sub-cohort 2, who received the EPI vaccination concomitantly with study vaccination with the Rotarix vaccine/placebo.
Time Frame: Within the 8-day (Days 0-7) follow-up periods following Dose 2 of the Rotarix vaccine/placebo
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 150 | 151
Participants
  Any Pain | 14 | 9
  Any Redness | 20 | 13
  Any Swelling | 13 | 6

10. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an unsolicited AE regardless of the intensity grade or relationship to vaccination.
Time Frame: Within the 31-day (Days 0-30) follow-up periods following any dose of the Rotarix vaccine or placebo
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1666 | 1667
Participants | 310 | 368

11. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, or result in disability/incapacity. Any = occurrence of an SAE regardless of the intensity grade or relationship to vaccination.
Time Frame: Throughout the entire study period (from Day 0 to Study End at Month 21)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 1666 | 1667
Participants | 183 | 246

12. Secondary Outcome: Number of Seroconverted Subjects for Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibodies
Description: A seroconverted subject was defined as a subject seronegative at baseline (Day 0) with the appearance of anti-RV IgA antibody concentration greater than or equal to (≥) 20 units per milliliter (U/mL) at the time point assessed. A seronegative subject was defined as a subject with anti-RV IgA antibody concentration lower than (<) 20 U/mL.
Time Frame: At Month 2 and at 12 months of age
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity Sub-cohort 1, which included subjects vaccinated with at least 1 dose of HRV vaccine/Placebo, complying with protocol, with EPI childhood vaccinations completed according to Chinese recommendations and available immunogenicity data at post sampling time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 257 | 254
Participants
  Anti-RV IgA - Month 2 | 192 | 9
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 246 | 252
  Anti-RV IgA - 12 months of age | 176 | 118

13. Secondary Outcome: Number of Seroconverted Subjects for Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibodies.
Description: as for outcome 12
Time Frame: At Month 2 and at 12 months of age
Population: Analysis was performed on the ATP cohort for immunogenicity Sub-cohort 2, which included subjects with OPV and Infanrix™ vaccines co-administered with the study vaccine, complying with protocol, with EPI childhood vaccinations completed according to Chinese recommendations and available immunogenicity data at post sampling time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 134 | 139
Participants
  Anti-RV IgA - Month 2 | 86 | 13
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 124 | 133
  Anti-RV IgA - 12 months of age | 62 | 29

14. Secondary Outcome: Number of Seroconverted Subjects for Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibodies.
Description: as for outcome 12
Time Frame: At Month 2 and at 12 months of age
Population: Analysis was performed on the ATP cohort for immunogenicity, which included eligible subjects in the ATP cohorts for immunogenicity sub-cohorts 1 and 2 seronegative for serum anti-rotavirus immunoglobulin A (IgA) antibodies at Day 0 and with availability immunogenicity data at pre and post sampling time-points.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 391 | 393
Participants
  Anti-RV IgA - Month 2 | 278 | 22
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 370 | 385
  Anti-RV IgA - 12 months of age | 238 | 147

15. Secondary Outcome: Number of Subjects Seropositive for Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibodies.
Description: A subject seropositive for anti-rotavirus (anti-RV) immunoglobulin A (IgA) antibodies was defined as a subject anti-RV IgA antibody concentration greater than or equal to (≥) the seropositivity cut-off of 20 units per milliliter (U/mL).
Time Frame: At Day 0, Month 2 and at 12 months of age
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 257 | 254
Participants
  Anti-RV IgA - Day 0 | 0 | 0
  Anti-RV IgA - Month 2 | 192 | 9
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 246 | 252
  Anti-RV IgA - 12 months of age | 176 | 118

16. Secondary Outcome: Number of Subjects Seropositive for Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibodies.
Description: as for outcome 15
Time Frame: At Day 0, Month 2 and at 12 months of age
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 134 | 139
Participants
  Anti-RV IgA - Day 0 | 0 | 0
  Anti-RV IgA - Month 2 | 86 | 13
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 124 | 133
  Anti-RV IgA - 12 months of age | 62 | 29

17. Secondary Outcome: Number of Subjects Seropositive for Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibodies.
Description: as for outcome 15
Time Frame: At Day 0, Month 2 and at 12 months of age
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 391 | 393
Participants
  Anti-RV IgA - Day 0 | 0 | 0
  Anti-RV IgA - Month 2 | 278 | 22
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 370 | 385
  Anti-RV IgA - 12 months of age | 238 | 147

18. Secondary Outcome: Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs), in units per milliliter (U/mL). The cut-off of the assay was the seropositivity cut-off (≥ 20 U/mL).
Time Frame: At Day 0, Month 2 and at 12 months of age
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 257 | 254
U/mL
  Anti-RV IgA - Day 0 | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL). | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL).
  Anti-RV IgA - Month 2 | 90.2 [73.3 to 111.1] | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL).
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 246 | 252
  Anti-RV IgA - 12 months of age | 66.5 [54.6 to 81.0] | 35.3 [29.3 to 42.5]

19. Secondary Outcome: Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibody Concentrations.
Description: as for outcome 18
Time Frame: At Day 0, Month 2 and at 12 months of age.
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 134 | 139
U/mL
  Anti-RV IgA - Day 0 | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL). | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL).
  Anti-RV IgA - Month 2 | 84.0 [58.9 to 119.8] | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL).
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 124 | 139
  Anti-RV IgA - 12 months of age | 31.3 [24.6 to 39.8] | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL).

20. Secondary Outcome: Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibody Concentrations.
Description: as for outcome 18
Time Frame: At Day 0, Month 2 and at 12 months of age
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Groups:
- Overall Study Arm: Subjects aged between and including 6 and 16 weeks at the time of first vaccination received 2 doses of Rotarix vaccine, liquid formulation, at Day 0 and at Month 1. As part of the routine childhood vaccination according to the Expanded Program of Immunization (EPI) recommendations in China, subjects in this group also received 3 doses of Infanrix vaccine and 3 doses of the oral poliovirus vaccine manufactured by the Institute of Medical Biology of the Chinese Academy of Medical Sciences (OPV). The Infanrix and the OPV vaccines were administered independently of (Sub-cohort 1) or concomitantly with (Sub-cohort 2) the Rotarix vaccine. When administered concomitantly, subjects received the 3 doses of Infanrix vaccine at Months 1, 2 and 3, and the 3 doses of the OPV vaccine at Day 0, Month 1 and Month 2. The Rotarix and OPV vaccines were administered orally; the Infanrix vaccine was administered intramuscularly in the left anterolateral thigh.
Arm/Group | Overall Study Arm | Placebo Group
Number analyzed (Participants) | 391 | 393
U/mL
  Anti-RV IgA - Day 0 | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL). | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL).
  Anti-RV IgA - Month 2 | 88.0 [73.4 to 105.6] | NA [NA to NA] — At this time-point, no subjects had an antibody concentration equal or above to the cut-off (20 U/mL).
  Anti-RV IgA - 12 months of age: number analyzed (Participants) | 370 | 385
  Anti-RV IgA - 12 months of age | 51.6 [44.1 to 60.5] | 27.4 [23.7 to 31.7]

21. Secondary Outcome: Number of Subjects Seroprotected Against Diphtheria and Tetanus
Description: A subject seroprotected against diphtheria/tetanus was defined as a subject with an anti-diphtheria (anti-D)/anti-tetanus (anti-T) antibody concentrations greater than or equal to (≥) 0.1 international units per milliliter (IU/mL). This outcome measure concerns solely subjects in Sub-cohort 2, who received the EPI vaccination concomitantly with study vaccination with the Rotarix vaccine/placebo
Time Frame: At Day 0 and at Month 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 133 | 139
Participants
  Anti-D at Day 0: number analyzed (Participants) | 133 | 138
  Anti-D at Day 0 | 1 | 1
  Anti-D at Month 4 | 133 | 139
  Anti-T at Day 0: number analyzed (Participants) | 133 | 138
  Anti-T at Day 0 | 0 | 1
  Anti-T at Month 4 | 133 | 139

22. Secondary Outcome: Anti-Diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) in international unit per milliliter (IU/mL). The cut-off of the assay was the seroprotection cut-off assay (≥ 0.1 IU/mL). This outcome measure concerns solely subjects in Sub-cohort 2, who received the EPI vaccination concomitantly with study vaccination with the Rotarix vaccine/placebo.
Time Frame: At Day 0 and at Month 4
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 133 | 139
IU/mL
  Anti-D at Day 0: number analyzed (Participants) | 133 | 138
  Anti-D at Day 0 | 0.051 [0.049 to 0.052] | 0.050 [0.050 to 0.051]
  Anti-D at Month 4 | 0.375 [0.326 to 0.432] | 0.334 [0.308 to 0.363]
  Anti-T at Day 0: number analyzed (Participants) | 133 | 138
  Anti-T at Day 0 | 0.050 [0.050 to 0.050] | 0.050 [0.050 to 0.051]
  Anti-T at Month 4 | 1.281 [1.253 to 1.309] | 1.343 [1.215 to 1.486]

23. Secondary Outcome: Number of Subjects Seroprotected Against Poliovirus Types 1, 2 and 3.
Description: A subject seroprotected against poliovirus types 1, 2 and 3 was defined as a subject with anti-poliovirus type 1 (anti-polio 1)/anti-polio 2/anti-polio 3 antibody titer greater than or equal to (≥) 8 estimated doses 50% (ED50). This outcome measure concerns solely subjects in Sub-cohort 2, who received the EPI vaccination concomitantly with study vaccination with the Rotarix vaccine/placebo (cf. population definition below).
Time Frame: At Day 0 and at Month 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 136 | 139
Participants
  Anti-polio 1 at Day 0 | 63 | 62
  Anti-polio 1 at Month 4 | 136 | 139
  Anti-polio 2 at Day 0 | 52 | 39
  Anti-polio 2 at Month 4 | 136 | 139
  Anti-polio 3 at Day 0 | 32 | 29
  Anti-polio 3 at Month 4 | 135 | 138

24. Secondary Outcome: Titers for Anti-poliovirus Type 1 (Anti-polio 1), Anti-polio 2 and Anti-polio 3 Antibodies
Description: Titers were expressed as geometric mean titers (GMTs). The cut-off of the assay was the seroprotection cut-off (≥ 8 estimated doses 50% [ED50] for anti-poliovirus type 1 [anti-polio 1]/anti-polio 2/anti-polio 3 antibodies. This outcome measure concerns solely subjects in Sub-cohort 2, who received the EPI vaccination concomitantly with study vaccination with the Rotarix vaccine/placebo.
Time Frame: At Day 0 and at Month 4
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 136 | 139
titers
  Anti-polio 1 at Day 0 | 8.9 [7.5 to 10.5] | 9.1 [7.6 to 11.0]
  Anti-polio 1 at Month 4 | 2101.1 [1734.8 to 2544.8] | 2259.4 [1844.4 to 2767.9]
  Anti-polio 2 at Day 0 | 7.6 [6.5 to 9.0] | 6.2 [5.4 to 7.1]
  Anti-polio 2 at Month 4 | 402.5 [334.8 to 483.9] | 425.1 [371.0 to 487.1]
  Anti-polio 3 at Day 0 | 5.6 [4.9 to 6.3] | 5.7 [4.9 to 6.6]
  Anti-polio 3 at Month 4 | 426.6 [342.7 to 531.0] | 360.3 [303.0 to 428.3]

25. Secondary Outcome: Number of Subjects Seropositive for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibodies.
Description: Antibody assessment was performed by enzyme-linked immunosorbent assay (ELISA). A subject seropositive for anti-PT/anti-FHA/anti-PRN antibodies was defined as a subject with an anti-PT/anti-FHA/anti-PRN antibody concentrations greater than or equal to (≥) 5 ELISA units per milliliter (EL.U/mL). This outcome measure concerns solely subjects in Sub-cohort 2, who received the EPI vaccination concomitantly with study vaccination with the Rotarix vaccine/placebo.
Time Frame: At Day 0 and at Month 4
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 133 | 139
Participants
  Anti-PT at Day 0: number analyzed (Participants) | 131 | 139
  Anti-PT at Day 0 | 43 | 34
  Anti-PT at Month 4 | 133 | 139
  Anti-FHA at Day 0: number analyzed (Participants) | 131 | 139
  Anti-FHA at Day 0 | 31 | 47
  Anti-FHA at Month 4 | 133 | 139
  Anti-PRN at Day 0: number analyzed (Participants) | 131 | 139
  Anti-PRN at Day 0 | 3 | 5
  Anti-PRN at Month 4 | 133 | 139

26. Secondary Outcome: Concentrations of Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibodies
Description: Antibody assessment was performed by enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA units per milliliter (EL.U/mL). The cut-off of the assay was the seropositivity cut-off (≥ 5 EL.U/mL) for all antibodies assessed (anti-PT, anti-FHA and anti-PRN). This outcome measure concerns solely subjects in Sub-cohort 2, who received the EPI vaccination concomitantly with study vaccination with the Rotarix vaccine/placebo.
Time Frame: At Day 0 and at Month 4
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 133 | 139
EL.U/mL
  Anti-PT at Day 0: number analyzed (Participants) | 131 | 139
  Anti-PT at Day 0 | 3.4 [3.1 to 3.7] | 3.2 [3.0 to 3.4]
  Anti-PT at Month 4 | 88.9 [84.9 to 93.2] | 90.5 [86.4 to 94.8]
  Anti-FHA at Day 0: number analyzed (Participants) | 131 | 139
  Anti-FHA at Day 0 | 3.1 [2.9 to 3.3] | 3.5 [3.2 to 3.8]
  Anti-FHA at Month 4 | 59.5 [55.8 to 63.5] | 65.8 [61.3 to 70.5]
  Anti-PRN at Day 0: number analyzed (Participants) | 131 | 139
  Anti-PRN at Day 0 | 2.6 [2.5 to 2.6] | 2.6 [2.5 to 2.7]
  Anti-PRN at Month 4 | 41.9 [37.6 to 46.5] | 50.8 [44.3 to 58.1]

ADVERSE EVENTS:
Time Frame: Solicited symptoms were collected during the 8-day (Days 0-7) post vaccination period. Unsolicited AEs were collected during the 31 day (Days 0-30) post vaccination. SAEs were collected throughout the entire study period (Months 0 to 21).
Description: One subject in the Placebo Group experienced an SAE assessed by the investigators as causally related to study vaccination (Diarrhoea).
Arm/Group | Rotarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 183/1666 | 246/1667
Other Adverse Events (participants affected / at risk) | 838/1666 | 880/1667
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=1666) | Placebo Group (N=1667)
Bronchitis (Infections and infestations) | 74 | 98
Bronchopneumonia (Infections and infestations) | 58 | 61
Enteritis (Gastrointestinal disorders) | 44 | 73
Pneumonia (Infections and infestations) | 14 | 14
Diarrhoea (Gastrointestinal disorders) | 4 | 11
Pharyngitis (Infections and infestations) | 2 | 8
Hand-foot-and-mouth disease (Infections and infestations) | 5 | 4
Tracheitis (Infections and infestations) | 4 | 4
Acute tonsillitis (Infections and infestations) | 5 | 2
Candidiasis (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 2 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 3
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Laryngitis (Infections and infestations) | 2 | 2
Diarrhoea infectious (Infections and infestations) | 1 | 2
Multi-organ failure (General disorders) | 1 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Convulsion (Nervous system disorders) | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 1
Febrile convulsion (Nervous system disorders) | 0 | 2
Gastroenteritis bacterial (Infections and infestations) | 0 | 2
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 2
Herpangina (Infections and infestations) | 1 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Intussusception (Gastrointestinal disorders) | 1 | 1
Pneumonia klebsiella (Infections and infestations) | 2 | 0
Thalassaemia beta (Congenital, familial and genetic disorders) | 2 | 0
Varicella (Infections and infestations) | 2 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Bacterial diarrhoea (Infections and infestations) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Central nervous system infection (Infections and infestations) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cortical dysplasia (Congenital, familial and genetic disorders) | 1 | 0
Death (General disorders) | 0 | 1
Deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shigella infection (Infections and infestations) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Thalassaemia (Congenital, familial and genetic disorders) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 16 | 26
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Bronchiolitis (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Rotarix Group (N=1666) | Placebo Group (N=1667)
Upper respiratory tract infection (Infections and infestations) | 119 | 124
Nasopharyngitis (Infections and infestations) | 103 | 123
Cough/runny nose (General disorders) | 313/1513 | 366/1514 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented, solely on subjects not part of Sub-cohort 2.
Diarrhoea (General disorders) | 127/1513 | 123/1514 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented, solely on subjects not part of Sub-cohort 2.
Irritability/Fussiness (General disorders) | 415/1513 | 448/1514 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented, solely on subjects not part of Sub-cohort 2.
Loss of appetite (General disorders) | 253/1513 | 250/1514 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented, solely on subjects not part of Sub-cohort 2.
Fever (GSK scale) (Axillary T >= 37.5°C) (General disorders) | 83/1513 | 104/1514 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented, solely on subjects not part of Sub-cohort 2.
Vomiting (General disorders) | 213/1513 | 232/1514 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented, solely on subjects not part of Sub-cohort 2.
Pain (General disorders) | 14/150 | 9/151 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.
Redness (General disorders) | 20/150 | 13/151 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.
Swelling (General disorders) | 13/150 | 6/151 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.
Drowsiness (General disorders) | 44/153 | 38/153 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.
Irritability/Fussiness (General disorders) | 56/153 | 52/153 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.
Loss of appetite (General disorders) | 43/153 | 32/153 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.
Fever - Chinese scale: Axillary T >= 37.1°C (General disorders) | 302/1513 | 313/1514 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented, solely on subjects not part of Sub-cohort 2.
Gastrointestinal symptoms (General disorders) | 43/153 | 38/153 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.
Fever - Chinese scale: Axillary T >= 37.1°C (General disorders) | 18/153 | 20/153 — The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the Rotarix™ vaccine or placebo administration documented only on subjects in sub-cohort 2, for whom results were available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.